CLINICAL TRIAL: NCT00095888
Title: A Phase II Trial Of Gemcitabine And Triapine In Refractory Metastatic Breast Cancer
Brief Title: 3-AP and Gemcitabine in Treating Patients With Refractory Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02632; MC0333; N01CM62205 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Gemcitabine

ARMS (1):
- Treatment (triapine, gemcitabine hydrochloride) (Experimental): Patients receive 3-AP (Triapine®) IV over 2 hours followed by gemcitabine IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: triapine; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of combining 3-AP with gemcitabine in treating patients who have refractory metastatic breast cancer. Drugs used in chemotherapy, such as 3-AP and gemcitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining 3-AP with gemcitabine may kill more tumor cells

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine antitumor activity of 3-AP (Triapine®) and gemcitabine by measuring tumor size in patients with refractory metastatic breast cancer.

Secondary I. Determine the safety and tolerability of this regimen in these patients. II. Determine the time to disease progression in patients treated with this regimen.

III. Determine the effect of multidrug resistance polymorphisms on pharmacokinetics and toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive 3-AP (Triapine®) IV over 2 hours followed by gemcitabine IV over 30 minutes on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 3 years after registration.

PROJECTED ACCRUAL: A total of 30-75 patients will be accrued for this study within 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer

  * Refractory metastatic disease
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Must have received 1, and only 1, prior chemotherapy regimen for metastatic disease
* Patients overexpressing HER2/neu antigen must have received a prior trastuzumab (Herceptin®)-containing regimen
* No known brain metastases
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-2
* At least 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* No uncontrolled congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No severe pulmonary disease requiring oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No glucose-6-phosphate dehydrogenase (G6PD) deficiency
* No other uncontrolled illness
* No active or ongoing infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to 3-AP (Triapine®) or other study agents
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy within the past 5 years
* See Disease Characteristics
* No concurrent immunotherapy
* No concurrent routine colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior gemcitabine for metastatic disease
* No other concurrent chemotherapy
* More than 4 weeks since prior hormonal therapy
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy
* Recovered from prior therapy
* No concurrent antiretroviral therapy for HIV-positive patients
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-10; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Confirmed response (complete or partial response) | Up to 6 months
  Ninety five percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Toxicities, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 3.0 | Up to 3 years
Time to progression | Time from registration to the time of progression, assessed up to 3 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Overall survival | Time from registration to death due to any cause, assessed up to 3 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Changes in tyrosyl radical and cell-cycle arrest on buccal mucosa | Pre-infusion, 2 and 4.5 hours post-infusion
Changes in R2 messenger ribonucleic acid (mRNA) on protein levels before and after treatment with triapine | Pre-infusion, 2 and 4.5 hours post-infusion
MDR polymorphism on tumor tissue | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: James Stewart, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States